CLINICAL TRIAL: NCT04500327
Title: An Exploratory Investigation of the Use of Drive App to Measure Sleep Parameters in Users of CPAP Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: DHT-20-04-01
Record Dates: First submitted 2020-05-26; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPAP users (Experimental): The Drive app will be used by CPAP users to identify any major issues with the usability and functionality of the app when used with CPAP therapy.
  Interventions: Other: Drive app; Device: Non contact motion sensor

INTERVENTIONS:
Other: Drive app — The Drive app will be used to monitor sleep metrics for users of CPAP therapy.
Device: Non contact motion sensor — The non contact motion sensor will be used as a reference to the Drive app i.e. Drive app overnight recordings will be compared to the non contact motion sensor overnight recordings.

SUMMARY:
The purpose of this study is to evaluate the usability and suitability of the Drive app (app under test) to measure sleep parameters during CPAP use.

This is a prospective, non-randomized, single arm exploratory study without blinding.

Current users of CPAP therapy will be recruited for this study and will be provided with a smartphone (app under test installed) and a non-contact motion sensor in their home environment. These devices will measure sleep metrics such as sleep stages and breathing metrics that may be associated with sleep disordered breathing. Usage and setup instructions will be provided for the study.

Participants will contribute up to 7 overnight recordings in the home environment and will complete daily questionnaires detailing their experience.

The study may be completed in two distinct phases, with an analysis performed after each phase. Each phase is expected to last up to six weeks with the overall study duration taking up to 12 months.

DETAILED DESCRIPTION:
The study may be completed in two distinct phases, with an analysis performed after each phase.

Phase 1 (Exploratory): A minimum of 10 and up to 12 participants will be recruited to identify any issues in using the app when used in conjunction with CPAP therapy (e.g. missed signals, inappropriate classification of breathing signals).

Phase 2 (Iterative Updates): Where changes to the algorithm or user interface are required, an additional 30 and up to 35 participants may be tested to provide design confidence. Conversely, if substantial issues are experienced and the time and effort required to address the issues is sufficiently large, the study may terminate before completion of phase 2.

Each phase is expected to last up to six weeks with the overall study duration taking up to 12 months.

Participants will be required to visit ResMed twice. The first visit will involve briefing of the study, consent form signatures, briefing on trial equipment and setup/usage instructions. The second (last) visit will involve going through the daily questionnaires with participants, collecting trial equipment and providing reimbursement for the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants willing to give written informed consent
* Participants who can read and comprehend English
* Participants who ≥ 18 years of age
* Participants established on CPAP therapy for the treatment of OSA for ≥ 6 months
* Participants who are able to set up the trial devices (ideally on a bedside table) with the following criteria:

  * Trial devices must be 10 cm higher than the mattress
  * Approx. 40 cm from the person's chest in bed
* Participants that have access to WI-FI in their home environment
* Participants who can trial the device for up to 7 nights
* *Participants who have been compliant (average of ≥4 hours of usage) to therapy for up to 7 nights of use

  * Note: the most recent consecutive 7 nights within the last 30 days

Exclusion Criteria:

* Participants using Bilevel flow generators
* Participants who are or may be pregnant, breastfeeding or within 6 weeks postpartum (which are known to cause significant sleep disruption)
* Participants with a preexisting lung disease/ condition that would predispose them to pneumothorax (for example: COPD, lung cancer; fibrosis of the lungs; recent (< 2years) case of pneumonia or lung infection; lung injury.
* Participants believed to be unsuitable for inclusion by the researcher
* *Participants using one of the following devices or Apps during the research period, or any other sleep tracking devices: SPlus, SleepScore app, SleepScore Max.

  * Note: If the participant uses the devices or apps above and they agree to delete/not use them during study period, they can be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Identify any failures when using the Drive app for users of CPAP therapy | 12 months (includes Phase 1 and Phase 2 and interim data analysis)
  This will be based on:
  1. Subjective data from daily questionnaires sent out to participants
  2. Comparison between Drive app data with the non contact motion sensor and CPAP data
  The questionnaire has yes/no questions and a likert scale (from 0-10) that participants fill in to indicate how representative each nights sleep hypnogram is. For e.g. if the participant was awake between 12am-1am but the app reports that the subject is in deep sleep, this will be captured in the questionnaire.
  Metrics including accuracy, correlation, total cohens kappa will be used for each signal recorded by the app which will be used to compare to the data from the reference devices.

SECONDARY OUTCOMES:
Evaluate usability of the Drive app | 12 months (includes Phase 1 and Phase 2 and interim data analysis)
  This will be based on subjective data from daily questionnaires sent out to participants.
  This data will be captured from comments by the participants in the daily questionnaires.
Compare subjective sleep quality data with data generated on the app. | 12 months (includes Phase 1 and Phase 2 and interim data analysis)
  This will be based on subjective data from daily questionnaires sent out to participants.
  The questionnaire has yes/no questions and a likert scale (from 0-10) that participants fill in to indicate how representative each nights sleep hypnogram is. For e.g. if the participant was awake between 12am-1am but the app reports that the subject is in deep sleep, this will be captured in the questionnaire.
Compare the Drive app sleep data to data from the reference devices. | 12 months (includes Phase 1 and Phase 2 and interim data analysis)
  Analyses will be performed to compare the Drive app data with the non contact motion sensor and CPAP device.
  Metrics including accuracy, correlation, total cohens kappa will be used for each signal recorded by the app which will be used to compare to the data from the reference devices.

CONTACTS AND LOCATIONS:
Locations (1):
- ResSleep, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No